CLINICAL TRIAL: NCT05817305
Title: Efficacy of an Exercise-based Secondary Prevention Program in Patients With Stable Cardiovascular Disease
Brief Title: Integrating Exercise Into Lifestyle of Cardiac Outpatients
Acronym: ITER
Status: Recruiting | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Giovanni Grazzi, MD, Professor, Università degli Studi di Ferrara
Other Study IDs: CSB-21-01
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Physical Inactivity; Aging; Quality of Life; Physician-Patient Relations
Keywords: Cardiovascular disease; Physical activity; Epidemiology; Cardiorespiratory fitness
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior; Motor Activity | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac outpatients: Patients with stable cardiovascular disease who have been referred to the service by their general practitioner or cardiologist
  Interventions: Other: Medical history and functional evaluation; Other: Health education

INTERVENTIONS:
Other: Medical history and functional evaluation — During each session, physical parameters are measured and data on medical history and physical activity are collected. To assess cardiorespiratory fitness, all patients complete a submaximal, moderate, and perceptually regulated treadmill walking test (1k-TWT). Patients unable to complete the test at a walking speed ≥ 3.0 km/h perform the test over 500m or 200m.
Other: Health education — Patients receive recommendations for risk factor management as well as continuous motivational counselling in order to develop and maintain a stable active lifestyle.

SUMMARY:
The purpose of the study is to investigate the long-term effects of a personalized physical activity program on exercise capacity and quality of life in patients with stable cardiovascular disease. The analysis also intends to evaluate the prognostic value of cardiovascular function estimated through a walking test (1km Treadmill Walking Test, 1k-TWT) in relation to survival, hospitalization, and medical costs. The program considers clinical, socio-economic, and behavioural aspects, psychological support, and risk factor control. Patients receive indications for carrying out a home training program based on the performance of moderate-intensity aerobic activity at least 3-4 days a week for at least 30-60 minutes a day. All patients are also encouraged to improve their daily habits by preferring a more active lifestyle both at home and at work.

DETAILED DESCRIPTION:
BACKGROUND: Physical activity and cardiorespiratory fitness are considered major markers of cardiovascular risk and core components of secondary prevention programs for cardiovascular diseases (CVD). The benefits of regular physical activity are well-recognized both for men and women and are inversely associated with mortality risk and the incidence of many chronic diseases. Despite the efforts of many health organizations to increase awareness of this evidence, physical inactivity and low cardiorespiratory fitness remain overlooked risk factors. Directly measured peak oxygen consumption (VO2peak) determined during maximal incremental cardiopulmonary exercise testing (CPX) is the gold standard objective measure of cardiorespiratory fitness. However, because of physical, financial, and time limitations, a direct determination is often not routinely assessed in clinical settings. Submaximal exercise testing can be a viable alternative to CPX. These tests are more practical for examining older adults or a large patient cohort. Also, they are helpful in defining functional limitations, setting up appropriate physical activity programs, and assessing the outcomes of pharmacological treatments.

RATIONALE AND OBJECTIVE OF THE STUDY: The benefits of regular physical activity are well-recognized both for men and women and are inversely associated with mortality risk and the incidence of many chronic diseases. The purpose of this observational registry is to evaluate the efficacy of an exercise-based secondary prevention program among male and female outpatients with stable cardiovascular disease.

DESCRIPTION OF THE FUNCTIONAL EVALUATION: During each session, information about weight, height, body mass index (BMI), blood pressure, cardiometabolic risk factors, and drug therapy in progress are registered. Physical activity habits are assessed using the Seven-Day Physical Activity Recall questionnaire. In addition, patients complete a sub-maximal test of 1km treadmill walking (1k-TWT), which is performed at a moderate intensity and adjusted according to the patient's perception of fatigue. Patients unable to complete the test at a walking speed ≥ 3.0 km/h can perform the test over 500m or 200m. Based on the results of the test, patients receive indications for the proper execution of a home training program, (i.e., at the same effort perceived in the test). The activity should be done at least 3-4 times per week, preferably every day, for at least 30-60 minutes. All patients are also encouraged to improve their daily habits by opting for a more active lifestyle at home and at work. Written informed consent is required from all participants at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* the presence of one or more previous cardiovascular events

Exclusion Criteria:

* Ejection fraction < 30%
* Chronic heart failure NYHA III-IV
* Severe aortic or mitral valvulopathy
* Severe physical or cognitive impairment
* Exercise-induced complex arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male and female outpatients with stable cardiovascular disease involved in an exercise-based secondary prevention program.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1997-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2047-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | From date of enrollment until the date of end of follow-up or date of death from any cause, whichever came first, assessed up to 12 years
  Association of all-cause mortality and cause-specific death with exercise capacity

SECONDARY OUTCOMES:
Hospitalization | From date of enrollment until the first hospitalization (any hospital admission is considered an event), assessed up to 12 years
  Association of cause-specific hospitalization with exercise capacity
Peak Oxygen Uptake (VO2peak) | From date of enrollment until the date of end of follow-up or date of death from any cause, whichever came first, assessed up to 12 years
  Measurement of cardiorespiratory fitness, reported as ml/kg/min and estimated through a moderate and perceptually regulated 1km treadmill walk test (1k-TWT) or through related short-forms (500m or 200m)
Leisure time physical activity levels | From date of enrollment until the date of end of follow-up or date of death from any cause, whichever came first, assessed up to 12 years
  Measurement of physical activity levels, reported as MET/h-week and estimated through the 7-day physical activity recall questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Mazzoni, Professor, Study Director — Università degli Studi di Ferrara; Giovanni Grazzi, Professor, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Center for Exercise Science and Sport, Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiaranda G, Myers J, Mazzoni G, Terranova F, Bernardi E, Grossi G, Codeca L, Conconi F, Grazzi G. Peak oxygen uptake prediction from a moderate, perceptually regulated, 1-km treadmill walk in male cardiac patients. J Cardiopulm Rehabil Prev. 2012 Sep-Oct;32(5):262-9. doi: 10.1097/HCR.0b013e3182663507. PMID 22936157
- [Background] Chiaranda G, Bernardi E, Codeca L, Conconi F, Myers J, Terranova F, Volpato S, Mazzoni G, Grazzi G. Treadmill walking speed and survival prediction in men with cardiovascular disease: a 10-year follow-up study. BMJ Open. 2013 Oct 25;3(10):e003446. doi: 10.1136/bmjopen-2013-003446. PMID 24163203
- [Background] Grazzi G, Myers J, Bernardi E, Terranova F, Grossi G, Codeca L, Volpato S, Conconi F, Mazzoni G, Chiaranda G. Association between VO(2) peak estimated by a 1-km treadmill walk and mortality. A 10-year follow-up study in patients with cardiovascular disease. Int J Cardiol. 2014 May 1;173(2):248-52. doi: 10.1016/j.ijcard.2014.02.039. Epub 2014 Feb 28. PMID 24630380
- [Background] Grazzi G, Mazzoni G, Myers J, Codeca L, Pasanisi G, Napoli N, Guerzoni F, Volpato S, Conconi F, Chiaranda G. Improved walking speed is associated with lower hospitalisation rates in patients in an exercise-based secondary prevention programme. Heart. 2016 Dec 1;102(23):1902-1908. doi: 10.1136/heartjnl-2015-309126. Epub 2016 Jul 7. PMID 27390367
- [Background] Uliari S, Myers J, Bernardi E, Chiaranda G, Conconi F, Terranova F, Mazzoni G, Grazzi G. Oxygen Uptake Attenuation at Ventilatory Threshold in Men With Coronary Artery Disease. J Cardiopulm Rehabil Prev. 2016 Jul-Aug;36(4):258-62. doi: 10.1097/HCR.0000000000000160. PMID 27120036
- [Background] Mandini S, Grazzi G, Mazzoni G, Myers J, Pasanisi G, Sassone B, Conconi F, Chiaranda G. A moderate 1-km treadmill walk predicts mortality in men with mid-range left ventricular dysfunction. Eur J Prev Cardiol. 2017 Oct;24(15):1670-1672. doi: 10.1177/2047487317722434. Epub 2017 Jul 21. No abstract available. PMID 28728484
- [Background] Grazzi G, Chiaranda G, Myers J, Pasanisi G, Lordi R, Conconi F, Mazzoni G. Outdoor Reproducibility of a 1-km Treadmill Walking Test to Predict Peak Oxygen Uptake in Cardiac Patients. J Cardiopulm Rehabil Prev. 2017 Sep;37(5):347-349. doi: 10.1097/HCR.0000000000000266. PMID 28671933
- [Background] Mazzoni G, Sassone B, Pasanisi G, Myers J, Mandini S, Volpato S, Conconi F, Chiaranda G, Grazzi G. A moderate 500-m treadmill walk for estimating peak oxygen uptake in men with NYHA class I-II heart failure and reduced left ventricular ejection fraction. BMC Cardiovasc Disord. 2018 Apr 16;18(1):67. doi: 10.1186/s12872-018-0801-9. PMID 29661150
- [Background] Mazzoni G, Chiaranda G, Myers J, Sassone B, Pasanisi G, Mandini S, Volpato S, Conconi F, Grazzi G. 500-meter and 1000-meter moderate walks equally assess cardiorespiratory fitness in male outpatients with cardiovascular diseases. J Sports Med Phys Fitness. 2018 Sep;58(9):1312-1317. doi: 10.23736/S0022-4707.17.07525-9. Epub 2017 Sep 29. PMID 28967238
- [Background] Grazzi G, Mazzoni G, Myers J, Codeca L, Pasanisi G, Mandini S, Piepoli M, Volpato S, Conconi F, Chiaranda G. Determining the best percent-predicted equation for estimated VO2 peak by a 1-km moderate perceptually-regulated treadmill walk to predict mortality in outpatients with cardiovascular disease. J Sci Med Sport. 2018 Mar;21(3):307-311. doi: 10.1016/j.jsams.2017.06.003. Epub 2017 Jun 8. PMID 28645496
- [Background] Grazzi G, Mazzoni G, Myers J, Caruso L, Sassone B, Pasanisi G, Guerzoni F, Napoli N, Pizzolato M, Zerbini V, Franchi M, Masotti S, Mandini S, Raisi A, Chiaranda G. Impact of Improvement in Walking Speed on Hospitalization and Mortality in Females with Cardiovascular Disease. J Clin Med. 2020 Jun 5;9(6):1755. doi: 10.3390/jcm9061755. PMID 32517001
- [Background] Mazzoni G, Myers J, Sassone B, Pasanisi G, Mandini S, Raisi A, Pizzolato M, Franchi M, Caruso L, Missiroli L, Chiaranda G, Grazzi G. A moderate 200-m walk test estimates peak oxygen uptake in elderly outpatients with cardiovascular disease. J Sports Med Phys Fitness. 2020 May;60(5):786-793. doi: 10.23736/S0022-4707.20.10387-6. PMID 32438791
- [Background] Bonnini S, Mazzoni G, Borghesi M, Chiaranda G, Myers J, Mandini S, Raisi A, Masotti S, Grazzi G. Improving walking speed reduces hospitalization costs in outpatients with cardiovascular disease. An analysis based on a multistrata non-parametric test. BMC Health Serv Res. 2020 Nov 17;20(1):1048. doi: 10.1186/s12913-020-05874-3. PMID 33203408
- [Background] Chiaranda G, Myers J, Arena R, Kaminsky L, Sassone B, Pasanisi G, Mandini S, Mazzoni G, Grazzi G. Prognostic comparison of the FRIEND and Wasserman/Hansen peak VO2 equations applied to a submaximal walking test in outpatients with cardiovascular disease. Eur J Prev Cardiol. 2021 Apr 23;28(3):287-292. doi: 10.1177/2047487319871728. Epub 2019 Aug 26. PMID 33891689
- [Background] Zerbini V, Raisi A, Myers J, Piva T, Lordi R, Chiaranda G, Mazzoni G, Grazzi G, Mandini S. Peak Oxygen Uptake Estimation From A Moderate 1-KM Treadmill Walk in Women With Cardiovascular Disease. J Cardiopulm Rehabil Prev. 2021 Nov 1;41(6):432-434. doi: 10.1097/HCR.0000000000000641. No abstract available. PMID 34727562
- [Background] Raisi A, Zerbini V, Myers J, Masotti S, Piva T, Lordi R, Chiaranda G, Grazzi G, Mazzoni G, Mandini S. Moderate walking speed and survival association across 23-years follow-up in female patients with cardiovascular disease. Int J Cardiol. 2023 Jan 15;371:371-376. doi: 10.1016/j.ijcard.2022.09.014. Epub 2022 Sep 9. PMID 36089160
- [Background] Raisi A, Piva T, Myers J, Lordi R, Zerbini V, Masotti S, Chiaranda G, Grazzi G, Mazzoni G, Mandini S. A Moderate Walking Test Predicts Survival in Women With Cardiovascular Disease. Am J Prev Med. 2023 Sep;65(3):497-504. doi: 10.1016/j.amepre.2023.02.025. Epub 2023 Mar 5. PMID 36871638
- [Derived] Raisi A, Bernardi E, Myers J, Piva T, Zerbini V, Masotti S, Menegatti E, Caruso L, Mazzoni G, Grazzi G, Mandini S. Change in Peak Oxygen Uptake Predicted by the Moderate 1-km Treadmill Walking Test After Walking Training in Outpatients With Cardiovascular Disease. J Cardiopulm Rehabil Prev. 2024 Mar 1;44(2):131-136. doi: 10.1097/HCR.0000000000000812. Epub 2023 Aug 25. PMID 37616588